CLINICAL TRIAL: NCT02293876
Title: Risk for Corneal Injury in Critically Ill Patients and Effect of Nursing Interventions for Its Prevention: Randomized Controlled Trial
Brief Title: Corneal Lesions in Intensive Care Unit (ICU) Clinical Trial for Proposing Interventions and Evaluating Outcomes of Nursing in the Adult Intensive Care Center Clinical Trial for Proposing Interventions and Evaluating Outcomes of Nursing in the Adult Intensive Care Center
Acronym: CORNEALPREV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Risoleta Tolentino Neves (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Andreza Werli Alvarenga, RN, MD, PhD, Hospital Risoleta Tolentino Neves
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: ICU CORNEAL ULCER 01
Record Dates: First submitted 2014-11-14; First posted 2014-11-18 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Keratitis; Corneal Ulcer
Keywords: Corneal Diseases; Corneal Ulcer; Nursing Diagnosis; Intensive Care Units; Nursing; Randomized Clinical Trial
MeSH Terms: conditions — Keratitis; Corneal Ulcer; Corneal Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Eye drop (Sham Comparator): Eye drop LACRIBELL® - two drops each eye, three times a day, after eye cleansing.
  Interventions: Device: LACRIBELL®
- Ocular gel (Sham Comparator): Ocular gel LIPOSIC® applied three times a day at the lower palpebra from medium line to the lateral border.
  Interventions: Device: LIPOSIC®
- Glad wrap (Sham Comparator): Occlusion of the orbital area with a Glad wrap, turning the area into a moisture chamber.
  Interventions: Device: Glad wrap
- Control group (No Intervention): Ocular cleansing three times a day.

INTERVENTIONS:
Device: LACRIBELL® — Hypromellose and dextran based eyedrop, used in the treatment of dry eye.
  Other Names: Eyedrop
  Arms: Eye drop
Device: LIPOSIC® — Carbomer and Sorbitol based gel, used in the treatment of dry eye.
  Other Names: Occular Gel
  Arms: Ocular gel
Device: Glad wrap — A clear plastic wrap occluding eye and orbital area, turning the space into a moisture chamber.
  Other Names: Polyethylene film
  Arms: Glad wrap

SUMMARY:
The purpose of the study is find out the better measure to achieve corneal protection in an Intensive Care Unit.

DETAILED DESCRIPTION:
Critically ill patients are at higher risk for corneal injury and the mechanisms responsible for ocular lubrication and protection can be compromised. However, the literature diverges on which is the best clinical practice for treatment. There is a scale for assessing the risk for corneal injury. Thus, the general objective of this study was to evaluate the risk for developing corneal injury in critically ill patients and the effectiveness of three types of interventions: eye gel, eyedrops and polyethylene film, compared to the control group in its prevention. The specific objectives were: verify the most effective intervention for the prevention of corneal injury from the available literature and provided by: eye gel, eyedrops and polyethylene film compared to the control group who received eye care through randomized controlled clinical trial. Patients and methods: This study was a randomized controlled trial to determine the best care for the prevention of corneal injury from those available on the market (eye drops, eye gel and polyethylene film), compared to a control group (eye care) in the period from 09/07/2013 to 03/15/2014 .

ELIGIBILITY:
Inclusion Criteria:

* Ramsay sedation scale 5 or 6
* Glasgow coma scale lower than 7
* Use of oxygen therapy by facial device above 6 liters per minute or mechanical ventilation
* Blink reflex less than 5 times per minute or ocular globe exposure

Exclusion Criteria:

* Less than 48 hours in Intensive Care Unit

Ages: 18 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Keratitis | Five days
  Presence of keratitis visible with a cobalt light ophthalmoscope and fluorescein eye drop.

CONTACTS AND LOCATIONS:
Overall Officials: Andreza Werli-Alvarenga, RN, MD, PhD, Principal Investigator — Hospital Risoleta Tolentino Neves
Locations (1):
- Hospital Risoleta Tolentino Neves, Belo Horizonte, Minas Gerais, Brazil